CLINICAL TRIAL: NCT00565474
Title: A Multicenter, Prospective, Double-blind, Randomized, Placebo-controlled, 6-month Study to Establish the Effect of Fluvastatin 40 mg (b.i.d.) in the Prevention of the Development of Vascular Graft Disease in de Novo Renal Transplant Patients
Brief Title: Evaluation of the Effect of Fluvastatin 40 mg (b.i.d.) in the Prevention of the Development of Vasculopathy of the Graft in de Novo Renal Transplant Patients Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LESTX-ES-01
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Graft Vasculopathy
Keywords: Renal transplantation; fluvastatin
MeSH Terms: interventions — Fluvastatin

ARMS (2):
- 1 (Active Comparator): fluvastatin 40mg b.i.d.
  Interventions: Drug: Fluvastatin
- 2 (Placebo Comparator): Placebo b.i.d.
  Interventions: Drug: Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin — Graft vasculopathy

SUMMARY:
Principal objective is to investigate if the treatment with fluvastatin can prevent the progression of vascular graft disease in de novo renal transplant patients.

ELIGIBILITY:
Inclusion criteria:

* Patients where the investigator expects to prescribe cyclosporine, mycophenolate mofetil and corticosteroids as base immunosuppressive therapy, regardless of their participation in the study.
* Man or woman aged from 17 to 70 years.
* Patients that receive a first or second renal transplant from a non-living donor
* Patients where allograft biopsies may be performed.
* Patients receiving an identical or compatible ABO graft.
* Patients willing to give their written informed consent to all study issues.
* Women with child-bearing potential should use a medically proven contraceptive method during the study.
* Patients able to meet all study requirements.

Exclusion criteria:

* Patients with pre-transplant cholesterol levels above 240 mg/dl (6.2 mmol/l).
* Positive cross-match of T cells or ABO incompatibility with the donor.
* Recipients of multiorgan transplant.
* Patients with diabetes mellitus.
* HIV seropositive or with surface antigen of Hepatitis B .
* Kidney from a donor aged over 65 years.
* Last panel of reactive antibody (PRA) above 50%.
* Women who plan to get pregnant within 12 months, or who are pregnant and/or nursing.
* Patients with a history of cancer in the previous 5 years, except for patients successfully treated with localized carcinoma of squamous or basal cells of the skin, or cervix cancer in situ treated adequately.
* Patients receiving an investigational drug in the 30 days prior to the transplant and/or who will receive an investigational/non-registered drug during the study, except for the use of erythropoietin-stimulating products
* Patients with myocardial infarction within the 6 months prior to the transplant, uncontrollable cardiac arrhythmia or another severe or unstable medical condition probably affecting the safety of the patient or the study objectives.
* Patients with alcohol dependence or drug abuse not solved, or signs of organic lesion caused by alcohol, mental dysfunction or other factors limiting their ability to fully cooperate with the study.
* Patients where it is planned to perform an induction treatment with preparations containing antilymphocyte antibodies (ALG, ATG or OKT-3).
* Patients scheduled to receive cyclosporine i.v. for over 48 hours.
* Patients with liver dysfunction (ALT or AST values or total bilirubin 2 times above the upper limit of the normal ranges of the laboratory values).
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2001-09; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To determine if treatment with fluvastatin can prevent the progression of vascular graft disease. The difference between the vascular intimal thickness measured on the baseline biopsy and the biopsy at the end of the study between the two treatment group | three Yrs

SECONDARY OUTCOMES:
24-hour creatinine and proteinuria values at 6 months post-transplant, graft survival and patient survival at 6 months, differences in lipid profile between the treatment groups, incidence of rejection episodes treated and documented by biopsy at 6 | Three yrs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigative Site, Barcelona, Spain

REFERENCES:
- [Result] Seron D, Oppenheimer F, Pallardo LM, Lauzurica R, Errasti P, Gomez-Huertas E, Bosmans JL, Sanchez-Plumed J, Romero R, Marques M, Fulladosa X, Moreso F. Fluvastatin in the prevention of renal transplant vasculopathy: results of a prospective, randomized, double-blind, placebo-controlled trial. Transplantation. 2008 Jul 15;86(1):82-7. doi: 10.1097/TP.0b013e318174428d. PMID 18622282